CLINICAL TRIAL: NCT05948033
Title: Phase I/II Study of CD70 Targeted CAR-T Cell Treatment in CD70 Positive Relapsed/Refractory Lymphoma
Brief Title: CD70 Targeted CAR-T Cells in CD70 Positive Relapsed/Refractory Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: UTC Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-081
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Lymphoma
Keywords: CD70; Relapsed/Refractory
MeSH Terms: conditions — Lymphoma; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD70-targeting CAR-T cells (Experimental): Enrolled participants will be given a preconditioning regimen consisted of fludarabine and cyclophosphamide before the infusion of CD70-CAR T cells.
  Enrolled patients in this arm will be administered CD70-CAR T cells in 3+3 based escalation manner.
  Interventions: Biological: CD70-targeting CAR-T cells

INTERVENTIONS:
Biological: CD70-targeting CAR-T cells — Dose escalation:
  Dose1 (1×10^6 cells/kg) ,Dose 2(3×10^6 cells/kg) ,Dose 3 (1×10^7 cells/kg)
  Doseexpansion: RP2D
  Drug: Fludarabine
  Intravenous fludarabine 25-30 mg/m^2/day on days 5, -4, and -3.
  Drug: Cyclophosphamide
  Intravenous cyclophosphamide 300-500 mg/m^2/day on days -5, -4, and -3.

SUMMARY:
In this single-center, single-arm,prospective, open-label, phase 1/2 study, the safety and efficacy of autologous CD70 targeted chimeric antigen receptor modified T (CAR-T) cell therapy will be evaluated in patients with CD70 antigen positive Relapsed/Refractory Lymphoma . In this clinical trial, at least 12 eligible patients in dose escalation period will be enrolled to receive 3 doses of CD70-CAR cell therapy according to the "3+3" principle. In dose expansion period, additional at most 21 eligible patients will be enrolled to receive CD70-CAR-T cell therapy at dose of recommended phase 2 dose(RP2D).

DETAILED DESCRIPTION:
CAR-T cell therapy has been identified as a breakthrough therapy in hematologic malignancies,especially anti-CD19 CAR-T cell therapy in the treatment of r/r B-NHL has achieved remarkable efficacy.However, relapse with CD19-negative tumor after treatment with anti-CD19 CAR-T cells has been reported in different types of B-cell lymphoid malignancies, with a percentage up to 38% in patients with non-Hodgkin lymphoma (NHL).At present, the CAR-T cell treatment for HL is mainly confined to CD30 antigen,with an objective response rate (ORR) only 38%~62%. Therefore, a more effective treatment strategy is needed for these patients.

CD70, the membrane-binding ligand of the CD27 (a tumor necrosis factor receptor superfamily), has been reported to mediate tumour cell proliferation and be expressed on the malignant cells of diffuse large B-cell lymphoma (DLBCL)，mantle cell lymphoma (MCL) and follicular lymphomas (FL), as well as Hodgkin lymphoma, etc,but rarely on normal B cells or T cells,indicating CD70 targeted treament has emerged as potentialnovel immunotherapeutic strategy.Preclinical study demonstrated CD70-CAR-T cells represent a new therapeutic option for the treatment of patients with CD19-negative recurrence of lymphoma.Based on the preclinical data, we conduct this clinical trial in order to test the the safety profiles and anti-tumor activities of CD70-CAR-T cells in vivo. In dose escalation period, at least 12 eligible patients will be enrolled and receive 3 doses of CD70-CAR-T cell therapy (1 × 10^6 cells/kg, 3 × 10^6 cells/kg, 1 × 10^7 cells/kg) according to the "3+3" principle. In dose expansion period, additional at most 21 eligible patients will be enrolled to receive CD70-CAR-T cell infusion at dose of RP2D, which is determined by data from dose escalation period, including occurrence of dose limiting toxicities(DLT), pharmacokinetics/pharmacodynamics, efficacy and other parameters, to furtherly evaluate the safety and efficacy profiles of CD70-CAR-T cell therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study had to meet all of the following criteria:

1. Age 18-75 (inclusive);
2. ECOG performance status ≤2 and Estimated life expectancy of more than 3 months;
3. Patients with histologically confirmed lymphoma including the following types defined by the World Health Organization(WHO) 2016:HL,Aggressive B-cell non-Hodgkin's lymphoma(Diffuse large B-cell lymphoma,High grade B-cell lymphoma,burkitt's lymphoma,Mantle cell lymph,Anaplastic large cell lymphoma, etc.) and Indolent lymphoma（Including but not limited to follicular lymphoma, marginal zone lymphoma, chronic lymphocytic leukemia, etc.）
4. Relapse after treatment with ≥2 lines systemic therapy for all the above disease types. Relapse disease is defined as disease progression after last regimen. Refractory disease is defined as no CR tofirst-line therapy:

   * PD as best response to first-line therapy, or
   * SD as best response after at least 4 cycles of first-line therapy (eg, 4 cycles of R- CHOP), or
   * PR as best response after at least 6 cycles and biopsy-proven residual disease or disease progression ≤ 6 months of therapy, or
   * Refractory post-autologous stem cell transplant (ASCT) i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy prove recurrence in relapsed individuals) ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy.
   * Individuals must have received adequate prior therapy.
5. CD70 antigen expression percentage ≥ 10%.
6. Successful leukapheresis assessment and preculture of T cells;
7. According to Lugano response criteria 2014, there should be at least one evaluable tumor focus. Evaluable tumor focus was defined as that with the longest diameter of intranodal focus > 1.5cm, the longest diameter of extranodal focus > 1.0cm assessed by computed tomography (CT) ormagnetic resonance imaging (MRI).
8. Functions of important organs meet the following requirements:ANC≥≥1×10^9/L; Platelet count ≥50×10^9/L; Hemoglobin ≥80 g/L;Serum AST and serum ALT, ≤3.0 x ULN (≤5 x ULN for patients with liver metastases); Total serum bilirubin ≤3.0 x ULN); Serum creatinine ≤1.5xULN ; Echocardiography showed left ventricular ejection fraction ≥50%.Pulmonary function: oxygen saturation of blood (SaO2) ≥92% in indoor air environment.
9. Toxicity from previous antitumor therapy ≤ grade 1 (according to CTCAE version 5.0) or to an acceptable level of inclusion/exclusion criteria (other toxicities such as alopecia and vitiligo considered by the investigator to pose no safety risk to the subject).
10. Pregnancy tests for women of childbearing age shall be negative;Both men and women agreed to use effective contraception during treatment and during the subsequent 1 year.
11. Ability to understand and sign a written informed consent documen.

Exclusion Criteria:

1. Subjects are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
2. Received cytotoxic chemicals, monoclonal antibodies, or immunotherapy within 4 weeks or 5 half-lives before enrollment;
3. Pregnant, lactating, or breastfeeding females;
4. Evidence of active uncontrolled viral, bacterial, or systemic fungal infection.
5. Known positive test result for human immunodeficiency virus (HIV) oracquired immune deficiency syndrome (AIDS);Active infection of hepatitis B virus (HBV), or hepatitis C virus (HCV);
6. History of allergy or intolerance to study drug components;
7. Prior organ allograft transplantations or allogeneic hematopoietic stem cell transplantation;
8. Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered.
9. Known brain metastases or active central nervous system(CNS) has been involved
10. Previous or concurrent cancer within 5 years prior to treatment start except for curatively treated cervical cancer in situ, non-melanoma skin cancer, local prostate cancer after radical surgery ;
11. Any serious underlying medical (eg, pulmonary, renal,hepatic,gastrointestinal, or neurological) or psychiatric condition or any issue that would limit compliance with study requirements;
12. Vaccination within 30 days of study enrollment;
13. Previously received targeting CD70 therapy;
14. Being participating any other trials or withdraw within 4 weeks;
15. Researchers believe that other reasons are not suitable for clinicaltrials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events（AEs） | Up to 12 months since the initiation of CD70-CAR-T cell therapy.
  AE is defined as any adverse medical event from the date of randomization to 12 months after CD70-CAR-T cells infusion. Among them, CRS and ICANS were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
Incidence of dose limiting toxicities (DLTs) | Up to 28 days since the initiation of CD70-CAR-T cell therapy
  DLT was defined as CD70-CAR-T cells-related events with onset within first 28 days following infusion:
  Thedevelopment of Grade (G) 3 or higher grade CRS lasting > 2 weeks; All G4 non-hematologic toxicities.
Maximum tolerated dose (MTD) | Up to 28 days since the initiation of CD70-CAR-T cell therapy
  MTD is defined as the highest dose level of less than or equal to 2 DLT among the 6 subjects finally determined.

SECONDARY OUTCOMES:
Number and copy number of CD70-CAR-T cells | Up to 3 years
  Number and copy number of CD70-CAR-T cells are evaluated by number in peripheral blood and tumor tissue.
Objective response rate (ORR) | Up to 3 years
  The incidence of complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or unevaluable (UE) as the best response to treatment assessed by investigators and based on the Lugano 2014.
  assessment criterion
Progression Free Survival (PFS) | Up to 3 years
  Progression Free Survival is defined as the time from the initiation of CD70-CAR-T cell therapy to documented disease progression or death.
Time to response (TTR) | Up to 3 years
  TTR is defined as the time from CD70-CAR-T cell infusion to first assessed CR or PR by investigators and based on the Lugano 2014 assessment criterion.
Duration of response (DOR) | Up to 3 years
  Duration of response is defined as the time from objective response until documented tumor progression among responders.
Overall Survival (OS) | Up to 3 years
  Overall Survival is defined as the time from the initiation of CD70-CAR-T cell therapy to documented disease progression or death.
Pharmacodynamics: Peak level of cytokines in serum (phase 1 and phase 2) | Up to 28 days since the initiation of CD70-CAR-T cell therapy
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α), C reactive protein (CRP), ferritin. Peak was defined as the maximum post-baseline level of the cytokine.

CONTACTS AND LOCATIONS:
Overall Officials: Yangbin Zhao, Ph.D, Study Director — UTC Therapeutics Inc.
Locations (1):
- China, Beijing, Biotherapeutic Department of Chinsese PLA Gereral Hospital, China

IPD SHARING:
Plan to Share IPD: No